CLINICAL TRIAL: NCT01549210
Title: Multicentre Prospective Observational Study for Identification of Determinants of Disability and Quality of Life in Patients With Gout.
Brief Title: Italian Observational Study Assessing the Impact of Gout on Patients Disability and Quality of Life
Acronym: KING
Status: Completed | Type: Observational
Sponsor: Italian Society for Rheumatology (Other)
Responsible Party: Principal Investigator, Carlo Alberto Scire, MD, PhD, Coordinator of the Epidemiology Unit - SIR, Italian Society for Rheumatology
Other Study IDs: SIR-2011\OSS001
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Gout
Keywords: gout; gouty arthritis
MeSH Terms: conditions — Gout; Arthritis, Gouty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study aims to identify which characteristics are associated with disability and poor quality of life in patients suffering from gout. This is a multicentre prospective observational study carried out in a cohort of Italian patients with gout. Subjects are randomly selected from a list of patients referred to each participant rheumatology clinic in the previous 2 years. Clinical evaluations are performed at baseline, at 6 and 12 months; data are retrieved about sociodemographic variables, life-styles, history of gout, comorbidities and patterns of treatment. At each visit patients complete questionnaires assessing disability and health-related quality of life. Preplanned analyses will be performed to investigate predictors of disability and poor quality of life in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gout
* Must be able to understand questionnaires

Exclusion Criteria:

* Diagnosis not validated by rheumatologist
* Not able to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referring to rheumatologic clinics
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Functional disability | 1 year
  Health Assessment Questionnaire Disability Index (HAQ-DI)

SECONDARY OUTCOMES:
Health-related quality of life | 1 year
  Short Form-36 Physical Summary Scale (SF-36 PCS)

OTHER OUTCOMES:
Short Form-36 Mental Summary Scale (SF-36 MCS) | 1 year
Serum uric acid levels | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlo A Scirè, MD, PhD, Principal Investigator — Epidemiology Unit - Italian Society for Rheumatology
Locations (1):
- Dept of Rheumatology - IRCCS San Matteo Foundation, Pavia, Pavia, Italy